CLINICAL TRIAL: NCT02767778
Title: A Multicentric, Prospective, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Effectiveness of Low-frequency Pulsed Electromagnetic Fields (ELF-MF) in Acute Ischemic Stroke
Brief Title: Low-frequency Pulsed Electromagnetic Fields (ELF-MF) as Treatment for Acute Ischemic Stroke
Acronym: I-NIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed positive results
Sponsor: Campus Bio-Medico University (Other)
Collaborators: Nuovo Ospedale Civile S.Agostino Estense (Other); San Raffaele University Hospital, Italy (Other); University Hospital of Ferrara (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); University of Rome Tor Vergata (Other); Ospedale Sant'Eugenio di Roma, Italy (Unknown)
Responsible Party: Principal Investigator, Di Lazzaro Vincenzo, Prof, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I-NIC
Record Dates: First submitted 2016-04-27; First posted 2016-05-10 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Acute; Ischemic Stroke
Keywords: Acute ischemic stroke; Neuroprotection; Extremely low frequency magnetic fields
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- REAL Pulsed ELF-MF stimulation (Experimental): Patients will receive REAL pulsed ELF-MF stimulation and the standard of care for acute ischemic stroke, according to current guidelines.
  Interventions: Device: REAL Pulsed ELF-MF stimulation
- SHAM Pulsed ELF-MF stimulation (Sham Comparator): Patients will receive SHAM pulsed ELF-MF stimulation and the standard of care for acute ischemic stroke, according to current guidelines.
  Interventions: Device: SHAM Pulsed ELF-MF stimulation

INTERVENTIONS:
Device: REAL Pulsed ELF-MF stimulation — Within 48 hours from the onset of the stroke, the enrolled patients will undergo to 120 min, daily, pulsed ELF-MF treatment for 5 consecutive days, during their hospital stay.Pulsed ELF-MF stimulation will be administrated by a rectangular, flexible coil, positioned upon the ischemic hemisphere and connected to the pulse generator (B-01; IGEA, Carpi, Italy) producing a single-pulsed signal at 75±2 Hz, with a pulse duration of 1.3 ms and a peak intensity of the magnetic field of 1.8±0.2 mT.
  Arms: REAL Pulsed ELF-MF stimulation
Device: SHAM Pulsed ELF-MF stimulation — SHAM pulsed ELF-MF stimulation will be administrated by a rectangular, flexible coil, positioned upon the ischemic hemisphere and connected to the pulse generator (B-01; IGEA, Carpi, Italy). The device for SHAM stimulation is identical and produces the same auditory sensation of the device for REAL stimulation but the SHAM device has no stimulating effect on the brain.
  Arms: SHAM Pulsed ELF-MF stimulation

SUMMARY:
The main purpose of this multicentric, prospective, randomized, placebo-controlled, double-blind study is the validation of pulsed ELF-MF stimulation as non-invasive and safe tool to promote recovery in acute ischemic stroke patients.

124 patients with acute ischemic stroke will be recruited and randomly assigned to real or sham group. Patients will be stimulated with pulsed ELF-MF (75 Hz, 1,8 mT), for 120 min daily, for 5 consecutive days, starting within 48 hours from the onset of stroke.

The primary outcome will consist of reduction of the expected infarct growth at MR measured in the subacute and chronic phase. Secondary outcomes will explore clinical effectiveness, safety and tolerability of pulsed ELF-MF in acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* first onset, mono-hemispheric ischemic stroke in the middle cerebral artery territory;
* onset of symptoms within 48 hours;
* National Institutes of Health Stroke Scale (NIHSS) score between 4 and 25;
* signed written informed consent.

Exclusion Criteria:

* acute intracranial hemorrhage;
* previous ischemic or hemorrhagic stroke;
* lacunar stroke, defined as not involving the cortex and < 2.0 cm if measured on MRI diffusion-weighted images;
* contraindications to transcranial magnetic stimulation such as implanted metallic parts of implanted electronic devices or other metal in body;
* historical modified Rankin Scale (mRS) >1;
* other serious or complex disease that may confound treatment assessment;
* women known to be pregnant, lactating or having a positive or indeterminate pregnancy test;
* current participation in another study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-04; Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Change in the volume of the ischemic lesion measured by MRI | Baseline and 45 days
  The effect of pulsed ELF-MF on ischemic lesion volume will be evaluated by MR at baseline (within 48 hours from the onset of the stroke), and after the 5-days ELF-MF exposure (after 7 and 45 days from the onset of the stroke).

SECONDARY OUTCOMES:
Change in NIHSS score | Baseline and 90 days
  Clinical evaluations will be performed by means of international well-validated scales (NIHSS) at baseline (within 48 hours from the onset of the stroke), and after the 5-days ELF-MF exposure (after 7, 45 and 90 days from the onset of the stroke). Clinical outcome measure is the change from baseline in NIHSS score measured at different follow-up after pulsed ELF-MF exposure.
Change in mRS score | Baseline and 90 days
  Clinical evaluations will be performed by means of international well-validated scales (mRS) at baseline (within 48 hours from the onset of the stroke), and after the 5-days ELF-MF exposure (after 7, 45 and 90 days from the onset of the stroke). Clinical outcome measure is the change from baseline in mRS score measured at different follow-up after pulsed ELF-MF exposure.
Change in Barthel Index score | Baseline and 90 days
  Clinical evaluations will be performed by means of international well-validated scales (Barthel Index) at baseline (within 48 hours from the onset of the stroke), and after the 5-days ELF-MF exposure (after 7, 45 and 90 days from the onset of the stroke). Clinical outcome measure is the change from baseline in Barthel Index scores measured at different follow-up after pulsed ELF-MF exposure.
Incidence of adverse events (AEs) and severe AEs (SAEs) that are related to treatment. | 90 days
  Safety will be assessed by measuring the incidence of AEs and SAEs throughout the stimulation period and along 3-months follow-up.
Number of participants with abnormal vital parameters. | 5 days
  During the pulsed ELF-MF stimulation, patients will be continuously monitored by multimodal monitor that simultaneously measures and displays the relevant vital parameters (respiratory rate, heart rate, blood pressure, pulse oximetry).
Change in NIHSS score during the 5-days ELF-MF exposure period. | 5 days
  Early neurological worsening will be evaluated by change in NIHSS score during the 5-days ELF-MF exposure period.
Number of participants with hemorrhagic transformation of ischemic lesion at MRI . | 7 days
Incidence of mortality | 90 days
  Safety will be assessed by measuring the incidence of mortality throughout the stimulation period and along 3-months follow-up.
Number of patients requiring to stop treatment sessions | 90 days
Incidence of discomfort during treatment sessions | 90 days
  Ad hoc questionnaire to detect any discomfort created by ELF-MF stimulation (e.g. nausea, headache, palpitations, anxiety, sweating) will be administered daily during the whole hospital stay and, after the discharge, at each outward control.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Di Lazzaro, MD, Study Director — Institute of Neurology, Campus Biomedico University
Locations (1):
- Institute of Neurology, Campus Biomedico University, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided